CLINICAL TRIAL: NCT02996097
Title: Fractional Laser Assisted Steroid Therapy vs Intralesional Steroids in the Treatment of Keloids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00082453
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- CO2 ablative laser plus intralesional triamcinolone acetonide (Experimental): A topical eutectic mixture of local anesthetics (EMLA) cream or tetracaine 7%/lidocaine 23% will be applied to the both treatment sites and after sufficient anesthesia is attained, one keloid will be treated with the fractional CO2 laser using standard protocol as practiced in our clinics followed by intralesional triamcinolone acetonide. One lesion would be treated with fractional CO2 ablative laser followed with intralesional triamcinolone acetonide at 4 weeks intervals
  Interventions: Device: The Lutronic electronic carbon dioxide (eCO2) Plus laser system; Drug: Intralesional Triamcinolone Acetonide
- Intralesional triamcinolone acetonide alone (Active Comparator): A topical EMLA cream or tetracaine 7%/lidocaine 23% will be applied to the both treatment sites and after sufficient anesthesia is attained, one keloid will be treated with the fractional CO2 laser using standard protocol as practiced in our clinics followed by intralesional triamcinolone acetonide. The other chosen lesion would be treated with intralesional triamcinolone acetonide alone at 4 week intervals.
  Interventions: Drug: Intralesional Triamcinolone Acetonide

INTERVENTIONS:
Device: The Lutronic electronic carbon dioxide (eCO2) Plus laser system — CO2 ablative laser plus intralesional triamcinolone acetonide A topical EMLA cream or tetracaine 7%/lidocaine 23% will be applied to the both treatment sites and after sufficient anesthesia is attained, one keloid will be treated with the fractional CO2 laser using standard protocol as practiced in our clinics followed by intralesional triamcinolone acetonide. One lesion would be treated with fractional CO2 ablative laser followed with intralesional triamcinolone acetonide at 4 weeks intervals
  Arms: CO2 ablative laser plus intralesional triamcinolone acetonide
Drug: Intralesional Triamcinolone Acetonide

SUMMARY:
The purpose of this study is to compare the effects of fractional carbon dioxide (CO2) laser therapy immediately followed by intralesional steroid therapy against intralesional steroid therapy alone for the treatment of keloids.

DETAILED DESCRIPTION:
Intralesional corticosteroids remain the gold standard treatment for keloids. However, more effective therapies are desperately desired. Ablative fractional laser (AFL) treatment facilitates delivery of intralesional steroid more deeply and uniformly into the skin by creating vertical channels. Recent studies have showed that fractional laser assisted steroid therapy can be effective in the treatment of keloids. However the studies are lacking in comparing this treatment modality to the gold standard of intralesional steroids.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 17 at the screening visit;
* The subject is healthy, as determined by the investigator based on a medical evaluation including medical history;
* The subject has at least two keloids of comparative size and texture located on the same general anatomic location (trunk or back);
* The subject is willing and able to comply with the requirements of the protocol. In particular, subject must adhere to the visits schedule and concomitant therapy. The subject is willing to comply with the 4 week washout period;
* The subject has understood and signed an Informed Consent Form approved by the Institutional Review Board (IRB) prior to any investigational procedure

Exclusion Criteria:

Any subject who is meeting one or more of the following exclusion criteria at the screening visit and/or at the baseline visit will not be included in this study:

* The subject has an underlying known disease, a surgical or medical condition that in the opinion of the investigator might put the subject at risk
* The subject is pregnant or breastfeeding at the time of enrollment or is planning to become pregnant at any point during the study period
* The subject has a past history of coagulopathy
* The subject has an underlying dermatological disease that in the opinion of the investigator could interfere with the study evaluations
* The subject has used prohibited topical or systemic treatments without sufficient protocol-defined wash-out period prior to Baseline (checked at Screening and Baseline) or is unwilling to refrain from use during the study
* The subject is treated with anticoagulants or antiplatelet therapies
* The subject has a known allergy or sensitivity to any local anesthetic drug (e.g. EMLA or tetracaine 7%/lidocaine 23%) or a local antiseptic planned to be used for the laser.
* The subject is in an exclusion period from a previous study or is participating in another clinical trial
* The subject is an adult under guardianship or is hospitalized in a public or private institution, or is deprived of freedom
* The subject is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginette Okoye, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Department of Dermatology, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lesions
Groups:
- CO2 Ablative Laser PLUS Intralesional Triamcinolone Acetonide: A topical eutectic mixture of local anesthetics (EMLA) cream or tetracaine 7%/lidocaine 23% will be applied to the both treatment sites and after sufficient anesthesia is attained, one keloid will be treated with the Lutronic electronic carbon dioxide (eCO2) Plus fractional CO2 laser using standard protocol as practiced in our clinics followed by intralesional triamcinolone acetonide at 4 weeks intervals.
- Intralesional Triamcinolone Acetonide Only: A topical eutectic mixture of local anesthetics (EMLA) cream or tetracaine 7%/lidocaine 23% will be applied to the both treatment sites and after sufficient anesthesia is attained, one keloid will be treated with intralesional triamcinolone acetonide only at 4 week intervals.
Period: Overall Study
Arm/Group | CO2 Ablative Laser PLUS Intralesional Triamcinolone Acetonide | Intralesional Triamcinolone Acetonide Only
Started | 30; 30 lesions | 30; 30 lesions
Per Protocol Population | 22; 22 lesions | 22; 22 lesions
Completed | 19; 19 lesions | 19; 19 lesions
Not Completed | 11; 11 lesions | 11; 11 lesions
Not completed — Lost to Follow-up | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All enrolled participants had two keloids on them, each keloid selected for an intervention arm of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Composite Observer Score for Patient and Observer Scar Assessment Scale (POSAS)
Description: Data from POSAS Observer Scale will be collected and reported to assess vascularity, pigmentation, thickness, relief, pliability, and surface area of the keloids chosen for the research study. Total score range: 6-60; Higher scores mean a worse outcome. Mean composite score of the final visit was compared to the mean baseline score.
Time Frame: Once every 4 weeks for 16 weeks
Population: Analyzed 19 participants who completed the study (5 visits) in addition to the 3 participants who completed 3 of 5 visits to provide enough data for this analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: lesions
Arm/Group | CO2 Ablative Laser PLUS Intralesional Triamcinolone Acetonide | Intralesional Triamcinolone Acetonide Only
Number analyzed (Participants) | 22 | 22
Number analyzed (lesions) | 22 | 22
score on a scale | -9.5 [-12.2 to -6] | -8.9 [-11.7 to -6]

2. Primary Outcome: Mean Change in Composite Patient Score for Patient and Observer Scar Assessment Scale (POSAS)
Description: as for outcome 1
Time Frame: Once every 4 weeks for 16 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: lesions
Arm/Group | CO2 Ablative Laser PLUS Intralesional Triamcinolone Acetonide | Intralesional Triamcinolone Acetonide Only
Number analyzed (Participants) | 22 | 22
Number analyzed (lesions) | 22 | 22
score on a scale | -22.6 [-28.5 to -16.7] | -18.8 [-24.5 to -13.2]

ADVERSE EVENTS:
Time Frame: 14 months
Groups:
- CO2 Ablative Laser +/- Intralesional Triamcinolone Acetonide: 2 keloids on each patient will be selected as treatment sites. A topical eutectic mixture of local anesthetics (EMLA) cream or tetracaine 7%/lidocaine 23% will be applied to the both treatment sites and after sufficient anesthesia is attained, one keloid will be treated with the Lutronic electronic carbon dioxide (eCO2) Plus fractional CO2 laser using standard protocol as practiced in our clinics followed by intralesional triamcinolone acetonide at 4 weeks intervals. The other keloid will be treated with intralesional triamcinolone acetonide only at 4 week intervals.
Arm/Group | CO2 Ablative Laser +/- Intralesional Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02996097/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02996097/SAP_001.pdf